CLINICAL TRIAL: NCT02980601
Title: The Use of Integra in Coverage of Radial Forearm Free Flap Donor Site Defect
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00031531; CCCWFU 99915A (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2016-11-29; First posted 2016-12-02 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Head and Neck Cancer
Keywords: Traumatic Defect; Chronic Wounds
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Integra and a Split Thickness Skin Graft (STSG) (Experimental): A sheet of Integra directly on the wound bed with subsequent removal of the overlying silicone sheet and immediate application of a 0.008mm STSG.
  Interventions: Device: Integra plus STSG; Procedure: STSG
- Split Thickness Skin Graft (STSG) (Active Comparator): reconstruction as dictated by the protocol. They will either receive 1) a 0
  Interventions: Procedure: STSG

INTERVENTIONS:
Device: Integra plus STSG — A sheet of Integra directly on the wound bed with subsequent removal of the overlying silicone sheet and immediate application of a 0.008mm STSG
  Arms: Integra and a Split Thickness Skin Graft (STSG)
Procedure: STSG — 0.012mm STSG

SUMMARY:
The purpose of this research study is to compare the forearm free flap of patients with a traditional split thickness skin graft and those repaired with Integra (a skin substitute that helps to provide wound closure) and a split thickness skin graft. The study team will be looking at the subject's satisfaction with how the skin graft site looks and how well the skin graft site is functioning.

DETAILED DESCRIPTION:
The radial forearm fasciocutaneous free flap (hereafter referred to as RFFF) was described more than 30 years ago as a fasciocutaneous flap for microsurgical transfer. It was soon after established as a safe and reliable flap for transfer of fascia and cutaneous tissue. Currently, it is used to repair any defect in which a relatively thin island of skin is needed with a fascial strength layer . While the flap itself is very reliable, it leaves a donor site that can be very unsightly and has multiple known complications including loss of pronation, pain, paresthesias, cold intolerance, and skin graft necrosis. The donor site is typically covered with a split thickness skin graft (hereafter referred to as STSG). In an effort to minimize these complications, several groups have described a technique of placing Integra© dermal substitute (hereafter referred to as Integra) underneath the STSG to provide a thicker support and decrease overall morbidity associated with the defect. These studies have shown success in decreasing overall morbidity including increasing range of motion and improving aesthetic quality of the donor site. However, the largest study to date has included only 29 subjects. Furthermore, these studies do not provide a comparative cohort of subjects repaired with a classic STSG to show effectiveness of this technique when compared to a classic repair. Our goal is to perform a prospective study comparing subjects repaired with a classic STSG and those repaired with one step Integra and STSG applied at the same time. These subjects will be evaluated for overall donor site aesthetic quality and functional outcome as described below.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who receive a radial forearm free flaps in the included time period, including subjects with head and neck cancer, traumatic defects, chronic wounds, or any other problems that require a radical forearm free flap for reconstruction.
* Have had a distal, anterograde fasciocutaneous flap
* Age ≥ 18 years
* Ability to understand and the willingness to sign an IRB-approved informed consent document.
* Smokers and tobacco users will be included in this study

Exclusion Criteria:

* Subjects who have had an osteocutaneous or musculocutaneous flap.
* Subjects who have a radial forearm flap with a proximal skin flap or subjects that receive a "reverse" radial forearm flap
* Pregnant women will be excluded due to the lack of clinical studies evaluating INTEGRA template in pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-08-18 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Molnar, MD, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Started | 6 | 4
Completed | 1 | 1
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 1
Not completed — Graft loss | 1 | 0
Not completed — Failed to sign consent | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG) | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Skin Graft Necrosis.
Description: Number of participants with skin graft necrosis.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
participants | 2 | 1

2. Primary Outcome: Vancouver Scar Scale
Description: The Vancouver Scar Scale will measure donor site aesethetic quality and it encompasses 4 separate outcomes to be objectively assessed. Each has been separately reported in the literature for each group in different papers as previously mentioned. We will compare the final score as well as scores within each outcome.On a scale of 1-13; with higher score denoting worse outcome.
Time Frame: 1 Year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Vancouver Scar Scale - Pigmentation
Description: Pigmentation will be measured on the Vancouver Scar Scale. On a scale of 0-2; higher score denoting worse outcome.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Vancouver Scar Scale - Vascularity
Description: Vascularity will be measured on the Vancouver Scar Scale. On a scale of 0-3; higher score denoting worse outcome.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Vancouver Scar Scale - Pliability
Description: Pliability will be measured on the Vancouver Scar Scale. On a scale of 1-5; higher score denoting worse outcome.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Vancouver Scar Scale - Height
Description: Height will be measured on the Vancouver Scar Scale. On a scale of 0-3; higher score denoting worse outcome.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Hand Strength -Lateral Pinch
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: Pre-op
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 19.4 (4.176123) | 21.25 (2.165064)

8. Primary Outcome: Hand Strength -Lateral Pinch
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 14.57142857 (4.655477353) | 16.8 (3.059411708)

9. Primary Outcome: Hand Strength -Lateral Pinch
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 15.8 (4.833218389) | 19.33333333 (2.494438258)

10. Primary Outcome: Hand Strength -Lateral Pinch
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: 1 year
Population: Data not recorded.
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Hand Strength - Grip
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: pre-op
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 72.4 (19.82523644) | 79.25 (16.02146997)

12. Primary Outcome: Hand Strength - Grip
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 58.14285714 (22.94358654) | 66.4 (21.81375713)

13. Primary Outcome: Hand Strength - Grip
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 66.4 (25.49195952) | 81.66666667 (16.49915823)

14. Primary Outcome: Hand Strength - Grip
Description: Functional outcomes will be measured by using strength dynamometers.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Hand Strength- Pincer
Description: Functional outcomes will be measured by using strength dynamometers
Time Frame: pre-op
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 13.4 (4.176122604) | 14.75 (3.561951712)

16. Primary Outcome: Hand Strength- Pincer
Description: Functional outcomes will be measured by using strength dynamometers
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 11 (5.318431563) | 12.2 (5.306599665)

17. Primary Outcome: Hand Strength- Pincer
Description: Functional outcomes will be measured by using strength dynamometers
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: Lbs
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
Lbs | 13.4 (4.079215611) | 16 (3.265986324)

18. Primary Outcome: Hand Strength- Pincer
Description: Functional outcomes will be measured by using strength dynamometers
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Wrist Range of Motion- Flexion
Description: Functional outcomes will be measured by using electric goniometers so as to standardize the measurements. Wrist flexion and wrist extension
Time Frame: pre-op
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
degrees | 72.83333333 (15.44254585) | 68 (16.02146997)

20. Primary Outcome: Wrist Range of Motion- Flexion
Description: as for outcome 19
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
degrees | 66.42857143 (13.55261854) | 69 (12)

21. Primary Outcome: Wrist Range of Motion- Flexion
Description: as for outcome 19
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
degrees | 59.8 (11.66876172) | 68.333333 (6.236095645)

22. Primary Outcome: Wrist Range of Motion- Flexion
Description: as for outcome 19
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Wrist Range of Motion- Extension
Description: as for outcome 19
Time Frame: pre-op
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
degrees | 57.33333333 (9.689627902) | 49.66666667 (7.758060325)

24. Primary Outcome: Wrist Range of Motion- Extension
Description: as for outcome 19
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
degrees | 45 (15.58387445) | 47.5 (13.78404875)

25. Primary Outcome: Wrist Range of Motion- Extension
Description: as for outcome 19
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
degrees | 59.4 (21.10544953) | 70 (8.498365856)

26. Primary Outcome: Wrist Range of Motion- Extension
Description: as for outcome 19
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Number of Participant With Tendon Exposure
Description: Tendon exposure identified clinically.
Time Frame: 6 month
Measure: Number; unit: participants
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
participants | 2 | 1

28. Primary Outcome: Rate of Tendon Exposure
Description: Tendon exposure identified clinically.
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Patient Scar Assessment- Paresthesia
Description: Presence of paresthesia on a 1-10 scale , higher score denote worse outcomes
Time Frame: 3 month
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Patient Scar Assessment- Paresthesia
Description: Presence of paresthesia on a 1-10 scale , higher score denote worse outcomes
Time Frame: 6 month
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: Patient Scar Assessment- Paresthesia
Description: Presence of paresthesia on a 1-10 scale , higher score denote worse outcomes
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

32. Primary Outcome: The Disabilities of the Arm, Shoulder and Hand (QuickDASH) Questionnaire)
Description: Functional outcome as measured by pre and post operative assessment on the QuickDASH scale. On a scale of 0-100; with higher score denotes worse outcome measure
Time Frame: pre-op
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: The Disabilities of the Arm, Shoulder and Hand (QuickDASH) Questionnaire)
Description: as for outcome 32
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
score on a scale | 27.43333333 (18.01894065) | 29.525 (23.13118836)

34. Primary Outcome: The Disabilities of the Arm, Shoulder and Hand (QuickDASH) Questionnaire)
Description: as for outcome 32
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
score on a scale | -3.636363636 (26.31264662) | -9.090909091 (16.62356686)

35. Primary Outcome: The Disabilities of the Arm, Shoulder and Hand (QuickDASH) Questionnaire)
Description: as for outcome 32
Time Frame: 1 year
Population: data not recorded for all subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 1 | 0
score on a scale | 5 (11.056672193748) |

36. Primary Outcome: Percent of Wound Contracture
Description: Planimetry Software will be used to measure and determine percentage of wound contracture
Time Frame: 3 month
Population: data not recorded
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

37. Primary Outcome: Percent of Wound Contracture
Description: Planimetry Software will be used to measure and determine percentage of wound contracture
Time Frame: 6 month
Population: data not recorded
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

38. Primary Outcome: Percent of Wound Contracture
Description: Planimetry Software will be used to measure and determine percentage of wound contracture
Time Frame: 1 year
Population: data not recorded
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

39. Primary Outcome: Skin Pliability
Description: Skin pliability will be measuredusing a Cutometer MPA 580. We plan to measure Pliability (Ua), Elasticity (Ue), Retraction (Ur). Viscoelasticity (Uv), and Extension (Uf).
Time Frame: 1 year
Population: Data not collected
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 0 | 0

40. Other Pre Specified Outcome: Patient Scar Assessment
Description: Total score (20-200). Higher scores denote worse outcomes.
Time Frame: 3 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
score on a scale | 86.14285714 (26.03529786) | 82.25 (27.72521416)

41. Other Pre Specified Outcome: Patient Scar Assessment
Description: Total score (20-200). Higher scores denote worse outcomes.
Time Frame: 6 month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
score on a scale | 89.8 (78.170071) | 65.5 (20.5)

42. Other Pre Specified Outcome: Patient Scar Assessment
Description: Total score (20-200). Higher scores denote worse outcomes.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
Number analyzed (Participants) | 6 | 4
score on a scale | 24.5 (3.5) | 28 (0)

ADVERSE EVENTS:
Time Frame: Data was collected during the 1 year of study activities.
Description: Definitions do not differ.
Arm/Group | Integra and a Split Thickness Skin Graft (STSG) | Split Thickness Skin Graft (STSG)
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integra and a Split Thickness Skin Graft (STSG) (N=6) | Split Thickness Skin Graft (STSG) (N=4)
Subject deceased (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT02980601/Prot_SAP_000.pdf